CLINICAL TRIAL: NCT00182793
Title: Phase II Study of Tandem Cycle Dose-Intense Chemotherapy of Melphalan and Carboplatin, Thiotepa and Cyclophosphamide (STMP V) ± Trastuzumab Followed by Helical Tomotherapy or Local Regional Radiation Therapy for Stage IV Metastatic and Stage IIIB/C Breast Cancer
Brief Title: Combination Chemotherapy With or Without Trastuzumab Followed By an Autologous Stem Cell Transplant and Radiation Therapy in Treating Patients With Stage III or Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05042; P30CA033572 (NIH); CDR0000442105 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; inflammatory breast cancer; male breast cancer; recurrent breast cancer; invasive ductal breast carcinoma with predominant intraductal component; invasive ductal breast carcinoma; medullary ductal breast carcinoma with lymphocytic infiltrate; mucinous ductal breast carcinoma; Paget disease of the breast with invasive ductal carcinoma; papillary ductal breast carcinoma; tubular ductal breast carcinoma; invasive lobular breast carcinoma with predominant in situ component; invasive lobular breast carcinoma; comedo ductal breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms; Breast Neoplasms, Male; Carcinoma, Ductal, Breast; Carcinoma, Lobular | interventions — Trastuzumab; Carboplatin; Cyclophosphamide; Melphalan; Thiotepa; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients undergo stem cell collection. Patients receive high-dose melphalan IV with or without trastuzumab (Herceptin®). One day later, patients undergo autologous peripheral blood stem cell (PBSC) transplantation. No more than 7 weeks later, patients proceed to course 2. After recover from high-dose chemotherapy and autologous PBSC transplantation, patients with stage IIIB or IIIC disease undergo radiotherapy to the chest wall and lymph nodes. Patients with stage IV disease undergo radiotherapy using helical tomotherapy or standard radiotherapy to oligometastatic sites.
  Interventions: Biological: trastuzumab; Drug: melphalan; Procedure: adjuvant therapy; Procedure: autologous-autologous tandem hematopoietic stem cell transplantation; Procedure: bone marrow ablation with stem cell support; Radiation: radiation therapy
- Arm II (Experimental): Patients undergo stem cell collection. Patients receive high-dose carboplatin, thiotepa, and cyclophosphamide IV continuously over 4 days followed by autologous PBSC transplantation. After recover from high-dose chemotherapy and autologous PBSC transplantation, patients with stage IIIB or IIIC disease undergo radiotherapy to the chest wall and lymph nodes. Patients with stage IV disease undergo radiotherapy using helical tomotherapy or standard radiotherapy to oligometastatic sites.
  Interventions: Drug: carboplatin; Drug: cyclophosphamide; Drug: thiotepa; Procedure: adjuvant therapy; Procedure: autologous-autologous tandem hematopoietic stem cell transplantation; Procedure: bone marrow ablation with stem cell support; Radiation: radiation therapy

INTERVENTIONS:
Biological: trastuzumab — Cycle 1: 6 mg/kg on day -2 from PBSC reinfusion Cycle 2: 6 mg/kg on day -7 from PBSC reinfusion
  Arms: Arm I
Drug: carboplatin — Cycle 2: 800 mg/m2/96 hours on days -7 to -3 from PBSC reinfusion
  Arms: Arm II
Drug: cyclophosphamide — Cycle 2: 6000 mg/m2/96 hours on days -7 to -3 from PBSC reinfusion
  Arms: Arm II
Drug: melphalan — Cycle 1: 150 mg/m2 on day -1 from PBSC reinfusion
  Arms: Arm I
Drug: thiotepa — Cycle 2: 500 mg/m2/96 hours on days -7 to -3 from PBSC reinfusion
  Arms: Arm II
Procedure: adjuvant therapy — Tandem high-dose chemotherapy comprising melphalan, carboplatin, thiotepa, and cyclophosphamide with or without trastuzumab (Herceptin®) followed by autologous peripheral blood stem cell transplantation and helical tomotherapy or loco-regional radiotherapy.
Procedure: autologous-autologous tandem hematopoietic stem cell transplantation — Tandem high-dose chemotherapy comprising melphalan, carboplatin, thiotepa, and cyclophosphamide with or without trastuzumab (Herceptin®) followed by autologous peripheral blood stem cell transplantation.
Procedure: bone marrow ablation with stem cell support — Tandem high-dose chemotherapy comprising melphalan, carboplatin, thiotepa, and cyclophosphamide with or without trastuzumab (Herceptin®) followed by autologous peripheral blood stem cell transplantation
Radiation: radiation therapy — After recovery from high-dose chemotherapy and autologous PBSC transplantation; patients with stage IIIB or IIIC disease undergo radiotherapy to the chest wall and lymph nodes. Treatment should be delivered daily M-F @ 180-200 cGY/day to a total of 4,500 to 5,040 cGy.
  Patients with stage IV disease undergo radiotherapy using helical tomotherapy or standard radiotherapy to oligometastatic sites. Treatment should be delivered daily @180-220 cGY/day to a total of 4,000-5,000 cGy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. An autologous stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy with or without trastuzumab followed by an autologous stem cell transplant and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy with or without trastuzumab followed by an autologous stem cell transplant and radiation therapy works in treating patients with stage III or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of tandem high-dose chemotherapy comprising melphalan, carboplatin, thiotepa, and cyclophosphamide with or without trastuzumab (Herceptin®) followed by autologous peripheral blood stem cell transplantation and helical tomotherapy or loco-regional radiotherapy in patients with high-risk stage IIIB, IIIC, or IV breast cancer.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: Patients undergo stem cell collection.

* Course 1: Patients receive high-dose melphalan IV with or without trastuzumab (Herceptin®). One day later, patients undergo autologous peripheral blood stem cell (PBSC) transplantation. No more than 7 weeks later, patients proceed to course 2.
* Course 2: Patients receive high-dose carboplatin, thiotepa, and cyclophosphamide IV continuously over 4 days followed by autologous PBSC transplantation.

After recover from high-dose chemotherapy and autologous PBSC transplantation, patients with stage IIIB or IIIC disease undergo radiotherapy to the chest wall and lymph nodes. Patients with stage IV disease undergo radiotherapy using helical tomotherapy or standard radiotherapy to oligometastatic sites.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer, meeting 1 of the following stage criteria:

  * Stage IIIB or IIIC disease, meeting both of the following criteria:

    * Must have received prior neoadjuvant or adjuvant therapy
    * Must have undergone lumpectomy or mastectomy
  * Stage IV disease, meeting all of the following criteria:

    * Only 1-3 organ sites with disease involvement after induction chemotherapy
    * Achieved at least a partial response after induction chemotherapy
    * No more than 3 lesions in the organ sites combined
* Inflammatory breast cancer allowed
* Completed chemotherapy, surgery, or radiotherapy for breast cancer within the past 6 months
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 65 and under

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* Karnofsky 80-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* SGOT or SGPT ≤ 2 times upper limit of normal
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine ≤ 1.2 mg/dL
* Creatinine clearance ≥ 70 mL/min

Cardiovascular

* LVEF ≥ 55% by MUGA or echocardiogram

Pulmonary

* FEV_1 ≥ 60% of predicted
* DLCO ≥ 60% of the lower limit of predicted value
* Oxygen saturation > 92% on room air

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No autoimmune disorders
* No immunosuppressive condition
* No other malignancy within the past 5 years

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy except trastuzumab (Herceptin®)

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to adjacent or involved sites of disease that would preclude study radiotherapy

Surgery

* See Disease Characteristics

Other

* No other concurrent anticancer therapy

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Somlo, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Patients undergo stem cell collection. Patients receive high-dose melphalan IV with or without trastuzumab (Herceptin®), one day later, patients undergo autologous peripheral blood stem cell (PBSC) transplantation, no more than 7 weeks later, patients proceed to course 2; OR Patients receive high-dose carboplatin, thiotepa, and cyclophosphamide IV continuously over 4 days followed by autologous PBSC transplantation. After recover from high-dose chemotherapy and autologous PBSC transplantation, patients with stage IIIB or IIIC disease undergo radiotherapy to the chest wall and lymph nodes. Patients with stage IV disease undergo radiotherapy using helical tomotherapy or standard radiotherapy to oligometastatic sites.
Period: Overall Study
Arm/Group | All Patients
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 47 [32 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: 5-Year Relapse-free Survival Rate
Description: Estimated using the product-limit method of Kaplan and Meier. Relapse defined as appearance of any new lesions during or after protocol treatment. Whenever possible, relapses should be documented histologically.
Time Frame: From time of initial PBPC rescue until death or disease recurrence (disease progression for patients with stage IV disease), whichever came first, up to 5 years post treatment
Population: Patients from this study were combined with patients from a follow-up study in which 27 patients from this study met the eligibility requirements for meta-analysis.
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 27
percentage of participants | 53 [23 to 77]

2. Primary Outcome: 5-Year Overall Survival Rate
Description: Estimated using the product-limit method of Kaplan and Meier. Patients who were still alive were censored at the date of last follow-up
Time Frame: From time of initial PBPC rescue until the date of death from any cause, assessed up to 5 years post treatment.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 27
percentage of participants | 75 [41 to 92]

ADVERSE EVENTS:
Time Frame: Adverse events took place over a period of 4 years, 3 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 24/32
Other Adverse Events (participants affected / at risk) | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=32)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Endocrine disorder (Endocrine disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (15)
Hemoglobin decreased (Blood and lymphatic system disorders) | 30 (53)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 24 (36)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Endocrine disorder (Endocrine disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 17 (22)
Anal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (11)
Diarrhea (Gastrointestinal disorders) | 26 (40)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 11 (14)
Dysphagia (Gastrointestinal disorders) | 6 (7)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 16 (21)
Enteritis (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 4 (4)
Gastritis (Gastrointestinal disorders) | 5 (6)
Gastrointestinal disorder (Gastrointestinal disorders) | 9 (13)
Gingival pain (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 6 (6)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 7 (8)
Nausea (Gastrointestinal disorders) | 27 (47)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 10 (11)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Rectal mucositis (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (32)
Chest pain (General disorders) | 3 (3)
Chills (General disorders) | 16 (23)
Edema limbs (General disorders) | 16 (25)
Fatigue (General disorders) | 26 (43)
Fever (General disorders) | 17 (21)
General symptom (General disorders) | 1 (1)
Injection site reaction (General disorders) | 14 (16)
Irritability (General disorders) | 1 (1)
Localized edema (General disorders) | 3 (4)
Pain (General disorders) | 12 (15)
Catheter related infection (Infections and infestations) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 7 (8)
Sinusitis (Infections and infestations) | 3 (3)
Skin infection (Infections and infestations) | 3 (3)
Upper aerodigestive tract infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Intraoperative gastrointestinal injury - Teeth (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 10 (12)
Alanine aminotransferase increased (Investigations) | 21 (33)
Alkaline phosphatase increased (Investigations) | 10 (12)
Aspartate aminotransferase increased (Investigations) | 23 (32)
Coagulopathy (Investigations) | 16 (24)
Hypercholesterolemia (Investigations) | 2 (2)
INR increased (Investigations) | 3 (3)
Leukocyte count decreased (Investigations) | 22 (40)
Leukopenia (Investigations) | 5 (10)
Lymphocyte count decreased (Investigations) | 5 (10)
Lymphopenia (Investigations) | 5 (9)
Neutrophil count decreased (Investigations) | 26 (48)
Platelet count decreased (Investigations) | 28 (50)
Serum cholesterol increased (Investigations) | 7 (9)
Weight gain (Investigations) | 5 (5)
Weight loss (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 23 (36)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 12 (16)
Blood glucose increased (Metabolism and nutrition disorders) | 23 (37)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (7)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (9)
Serum albumin decreased (Metabolism and nutrition disorders) | 22 (38)
Serum calcium decreased (Metabolism and nutrition disorders) | 14 (22)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 16 (22)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 17 (20)
Serum potassium decreased (Metabolism and nutrition disorders) | 17 (23)
Serum sodium decreased (Metabolism and nutrition disorders) | 19 (21)
Serum triglycerides increased (Metabolism and nutrition disorders) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (11)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 10 (11)
Headache (Nervous system disorders) | 20 (33)
Neurological disorder NOS (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (12)
Sinus pain (Nervous system disorders) | 3 (3)
Taste alteration (Nervous system disorders) | 8 (10)
Tremor (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 13 (17)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 7 (8)
Insomnia (Psychiatric disorders) | 12 (13)
Personality change (Psychiatric disorders) | 1 (2)
Psychosis (Psychiatric disorders) | 2 (2)
Cystitis (Renal and urinary disorders) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 5 (6)
Renal failure (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 3 (6)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (15)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (16)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 10 (11)
Skin disorder (Skin and subcutaneous tissue disorders) | 4 (7)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 6 (9)
Hemorrhage (Vascular disorders) | 2 (3)
Hot flashes (Vascular disorders) | 7 (10)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 21 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes